CLINICAL TRIAL: NCT02005744
Title: A Pharmacokinetic Study of CKD-501 in Patients With Impaired Hepatic Function Compared With Normal Hepatic Function
Brief Title: A Pharmacokinetic Study of CKD-501 in Patients With Impaired Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 19HI13018
Record Dates: First submitted 2013-12-04; First posted 2013-12-09 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2014-05

CONDITIONS: Liver Dysfunction
Keywords: CKD-501
MeSH Terms: conditions — Liver Diseases | interventions — lobeglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Child Pugh A (Experimental): CKD-501 will be administered to patients who are included Child Pugh A
  Interventions: Drug: CKD-501
- Child Pugh B (Experimental): CKD-501 will be administered to patients who are included Child Pugh B
  Interventions: Drug: CKD-501
- Subject who are matched Child Pugh A (Experimental): CKD-501 will be administered to the Subjects who are matched Child Pugh A
  Interventions: Drug: CKD-501
- Subject who are matched Child Pugh B (Experimental): CKD-501 will be administered to the subjects who are matched Child Pugh B
  Interventions: Drug: CKD-501

INTERVENTIONS:
Drug: CKD-501 — CKD-501 0.5mg, PO(per oral), once
  Other Names: Lobeglitazone

SUMMARY:
The purpose of this study is to evaluate pharmacokinetics of CKD-501 in patients with impaired hepatic function compared with normal hepatic function.

DETAILED DESCRIPTION:
A Phase 1, Non-randomized, Open, Parallel-Group study.

ELIGIBILITY:
A. Inclusion Criteria

[The subjects with impaired hepatic function]

1. The subjects who are 19 to 64 years old
2. The subjects with stable hepatic disease and impaired hepatic function as Child-Pugh A or B
3. Body Weight ≥ 55kg
4. If females, Negative for pregnancy test at the screening and pre dose of Day 1
5. The subjects who agreed with performing contraception during the study
6. The subjects who agreed with written informed consent

[The subjects with normal hepatic function]

1. The subjects who are 19 to 64 years old
2. The subjects who are matched impaired hepatic function by gender, age(± 5years) and body weight(± 10kg)
3. If females, Negative for pregnancy test at the screening and pre dose of Day 1
4. The subjects who agreed with performing contraception during the study
5. The subjects who agreed with written informed consent

B. exclusion criteria

[The subjects with impaired hepatic function]

1. The subjects with impaired hepatic function as Child-Pugh C
2. The subjects had a portosystemic shunt surgery
3. The subjects had a liver transplantation or unsuitable for the study by the investigator's judgement(for examples, hepatic encephalopathy grade 3 or 4, stroke, heart failure, cancer etc.) but The subject is eligible to participate if had not chemotherapy or radiofrequency ablation therapy within 6months)
4. The subjects have a gastrointestinal disease or surgery which can be effected in absorption of Investigational product
5. The subjects who took drugs or medicine which can be effected in metabolism of Cytochrome P450 within 14days prior to Day 1
6. Positive for anti-HIV Ab or venereal disease research laboratory etc.

[The subjects with normal hepatic function]

1. The subjects with liver disease or abnormal Laboratory test(Asparate transaminase >1.25 fold of upper normal limit, Alanine transaminase>1.25 fold of upper normal limit, Total bilirubin >1.5 fold of upper normal limit)
2. The subjects have a gastrointestinal disease or surgery which can be effected in absorption of Investigational product
3. Estimated Glomerular filtration rate < 60 mL/min/1.73m2 by Modification of Diet in Renal Disease formula
4. Positive for HBsAg, anti-Hepatitis C virus Ab, anti-HIV Ab or venereal disease research laboratory
5. The subjects with high blood pressure or low blood pressure(systolic blood pressure >150mmHg or <100mmHg, diastolic blood pressure>90mmHg or <60mmHg)
6. The subjects who took drugs or medicine which can be effected in metabolism of Cytochrome P450 within 14days prior to Day 1 etc.

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2014-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration(last) and Cmax of CKD-501 | 0 to 48 hours
  Sampling timepoint(hours)
  : 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48

SECONDARY OUTCOMES:
Tmax, Area Under the Concentration(inf), T1/2 and Clearance/F of CKD-501 and its metabolite | 0 to 48 hours
  Sampling timepoint(hours)
  : 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48
Fraction Unbound of CKD-501 and its metabolite | 1 and 8 hours
  sampling timepoint(hours)
  : 1, 8
Area Under the Concentration(last) and Cmax of the metabolite | o to 48 hours
  sampling timepoint(hours)
  : 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48
Metabolic ratio(metabolite/CKD-501) | 0 to 48 hours
  sampling timepoint(hours)
  : 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48

OTHER OUTCOMES:
Vital signs | up to 8 days
Physical examination | up to 8 days
Laboratory tests | up to 8 days
Adverse events | up to 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Min Soo Park, Ph.D. M.D, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University Severance Hospital, Soeul, South Korea